CLINICAL TRIAL: NCT00201630
Title: Randomized, Open-Labeled Study of Prophylactic Vs. Therapeutic Use of Uroxatrol to Determine Improvements in Urinary Morbidity Following Men Undergoing Prostate Brachytherapy
Brief Title: Prophylactic Vs. Therapeutic Use of Uroxatrol in Men Undergoing Brachytherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Prostate Institute (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; cancer; Brachytherapy; Alpha Blocker
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — alfuzosin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Uroxatrol (drug)

SUMMARY:
To asess the efficacy of Uroxatrol, an alpha blocker in men undergoing prostate brachytherapy to treat prostate cancer, and whether the use of Uroxatrol in advance of the brachytherapy is better or not than starting it on the day of surgery.

DETAILED DESCRIPTION:
Prostate brachytherapy is an increasingly popular method of treating clinically localized prostate cancer. The major morbidity of this procedure is obstructive and irritative voiding symptoms. The risk of urinary retention in published series is 10-15%. Voiding symptoms persist up to 1 year following this procedure.

The primary experience in treating obstructive and irritative voiding symptoms is in men with benign prostatic hyperplasia (BPH). In patients with moderate to severe voiding symptomatology, based in the American Urological Association (AUA) Symptom Score Index, medical treatment with alpha antagonists has become commonplace. The use of alpha antagonists is based upon the reduction of smooth muscle tone in both the prostate gland and urinary bladder neck by inhibition of alpha1 adrenoceptor, resulting in relaxation of bladder outlet obstruction and increased urinary flow.

Alfuzosin hydrochloride was approved by the FDA for treatment of the signs and symptoms of BPH in 2003. Alfuzosin differs from other  1-adrenergic receptor blockers by the absences of a piperidine moiety and the presence of a diaminopropyl spacer, which confers alfuzosin with specific biochemical properties. Affinity studies on human-cloned  1 receptor subtypes show that alfuzosin, like terazosin and doxazosin, is devoid of significant receptor subtype selectivity. In isolated human tissues, however, alfuzosin displays the highest selectivity ratio for the prostate over the vascular tissue (ratio, 544) compared with tamsulosin (90), doxazosin (51), and terazosin (19).

Prostate cancer is the most common malignancy in men. One of the most common treatments of prostate cancer is prostate brachytherapy, or radioactive seed implantation. All patients are affected by obstructive and irritative voiding symptoms to various degrees following this procedure due to edema and inflammation induced by trauma and radiation. Many physicians routinely treat obstructive and irritative voiding symptoms following prostate brachytherapy with alpha-blockers. Patients presenting with clinically localized prostate cancer may elect permanent prostate brachytherapy as definitive therapy. The efficacy of such therapy matches that of radical prostatectomy or external beam radiation. Many patients select brachytherapy since it is a single treatment session that is considered minor surgery. Most patients are discharged the same day and they may resume their normal physical activities without restriction almost immediately.

However, the trauma of the needle sticks through the perineum coupled with the effects of the radiation can cause a prostatitis with symptoms similar to irritable bladder or benign prostatic hypertrophy. These symptoms can have considerable impact on the quality of life of the patient and many are medicated with alpha-blockers.

Several studies have attempted to define how best to predict for and treat these symptoms. However, the incidence and severity of these symptoms is difficult to predict. The prophylactic use of alpha-blockers may better control these symptoms in some men undergoing prostate brachytherapy. The aim of this study is to compare outcomes of urinary morbidity following prostate brachytherapy between patients treated with alfuzosin prior to implantation and patients treated following implantation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Informed consent must be obtained. 2) Men of any age 3) Diagnosis of prostate cancer that is clinically localized 4) Patients must be eligible for permanent prostate brachytherapy either alone or with combination of other treatments (i.e. External beam radiation or hormonal therapy)

Exclusion Criteria:

* Refusal to participate in the study
* Prior use of alpha-blocker or anti-cholinergic medication in the treatment of prostate hypertrophy.
* Contraindication to using an alpha-blocker

Min Age: 0 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2005-09; Study Completion 2005-09

PRIMARY OUTCOMES:
IPSS and sexual function QOL life

SECONDARY OUTCOMES:
Safety and tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Louis Potters, MD, Study Chair — New York Prostate Institue
Locations (1):
- New York Prostate Institute, Oceanside, New York, United States

REFERENCES:
- [Background] Lefevre-Borg F, O'Connor SE, Schoemaker H, Hicks PE, Lechaire J, Gautier E, Pierre F, Pimoule C, Manoury P, Langer SZ. Alfuzosin, a selective alpha 1-adrenoceptor antagonist in the lower urinary tract. Br J Pharmacol. 1993 Aug;109(4):1282-9. doi: 10.1111/j.1476-5381.1993.tb13762.x. PMID 8104650
- See also: New York Prostate Institute web site — http://www.nyprostate.org